CLINICAL TRIAL: NCT04756596
Title: Development and Validation of a Web-based Digital Distance Visual Acuity Test
Brief Title: A Web-based Digital Distance Visual Acuity Test
Acronym: DDVIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Democritus University of Thrace (Other)
Collaborators: University of Thessaly (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Professor (Associate) of Democritus University of Thrace, Democritus University of Thrace
Other Study IDs: ES1/Th6/21-1-2021
Record Dates: First submitted 2021-02-12; First posted 2021-02-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Refractive Errors; Low Vision; Vision Disorders
Keywords: web application; distance visual acuity; smart features; face detection; text calibration
MeSH Terms: conditions — Refractive Errors; Vision, Low; Vision Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: 70 patients with normal vision (NVG) 30 patients with low vision (LVG) These patients will be tested on the DDVIT
  Interventions: Diagnostic Test: DDVIT testing; Diagnostic Test: ETDRS testing

INTERVENTIONS:
Diagnostic Test: DDVIT testing — One randomly selected eye will be included for each study participant. Participants respond to the DDVIT test in standard environmental lighting conditions at 4 m viewing distance. Visual acuity will be evaluated.
Diagnostic Test: ETDRS testing — The same eye is included for each study participant. Participants respond to the standard ETDRS chart of our Ophthalmology Department in standard environmental lighting conditions at 4 m viewing distance. Visual acuity will be evaluated.

SUMMARY:
Primary objective of this study is the development and validation of a web-based application for the examination of the distance visual acuity of normal- and low-vision patients.

DETAILED DESCRIPTION:
Present study aims to develop and validate a web-based digital distance visual acuity test (Democritus Distance Vision Test - DDVIT). DDVIT is an application, which will be easily accessed through a simple internet connection. This application will provide the possibility of a simple but reliable examination of patients, establishing a commonly accepted way of measuring the distance visual acuity among rural doctors, general practitioners and ophthalmologists.

Specifically, present study aims to develop a new online distance visual acuity test (DDVIT) according to the standards of the Early Treatment Diabetic Retinopathy Study (ETDRS) test and to evaluate the level of agreement between the two visual acuity tests, as well as the test-retest reliability of the online DDVIT visual acuity test.

The first part of the study is the development of the online visual acuity test (letters, numbers, symbols) including the following smart features:

1. Adjustment of the font size according to the size of the computer screen used for the examination
2. Real time calculation of the patient-screen distance through a face detection system
3. Automatic calculation of the reading time of each line (each logMAR)
4. Entering the number of patient's reading errors for each line
5. Automatic calculation of the visual acuity in the following score units:

   * Number of Letters (max 85)
   * Visual Acuity Score (max 100)
   * logMAR
   * Decimal
   * Snellen Fraction

The calculation of various reading parameters resulting from the aforementioned features (visual acuity score in different units, reading duration (in sec) and number of errors for each slide (line), patient-screen distance for each slide) will be performed after the end of the examination. Except for the html format, a file in the format of Microsoft Excel and Pdf are also generated.

The second part of this study is the clinical validation of the DDVIT visual acuity test. In this part, the reading acuity measured with the DDVIT and ETDRS test are compared.

All the comparisons will take place in two groups: a) a Normal Vision Group (NVG), and b) a Low Vision Group (LVG) in order to estimate the visual acuity in a population with a wide range of vision.

ELIGIBILITY:
Inclusion Criteria:

* Patients of our outpatient ophthalmology clinic
* Age between 18 to 75 years

Exclusion Criteria:

* Dyslexia
* Attention-deficiency
* Former diagnosis of mental and/or psychiatric diseases
* Inability to cooperate

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Normal- and low-sighted participants aged 18 to 75 years.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Distance visual acuity using DDVIT vision test | 4 months
  The distance visual acuity of the one randomly selected eye of each participant will be evaluated by the examiner using DDVIT vision test.
Distance visual acuity using ETDRS vision test | 4 months
  The distance visual acuity of the same eye of each participant will be evaluated by the same examiner using the web-based ETDRS vision test under the same predetermined environmental lighting conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, MD, PhD, Study Chair — Department of Ophthalmology, University Hospital of Alexandroupolis, Alexandroupolis, Greece
Locations (2):
- Greece (2):
  - Department of Ophthalmology, University Hospital of Alexandroupolis, Alexandroupoli, Evros
  - Department of Computer Science and Biomedical Informatics, University of Thessaly, Lamía, Thessaly

IPD SHARING:
Plan to Share IPD: Undecided